CLINICAL TRIAL: NCT05673499
Title: International Study of Cerebral Oxygenation and Electrical Activity During Major Neonatal Surgery
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 22-019679
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Congenital Disorders; Cerebral Desaturation; Neonatal Surgery
Keywords: Electroencephalography; Near-infrared spectroscopy
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants: Infant subjects ≤ 60 weeks post-menstrual age who are undergoing surgery for congenital malformations
  Interventions: Device: NIRS/EEG monitoring

INTERVENTIONS:
Device: NIRS/EEG monitoring — The study intervention will be monitoring NIRS and EEG for one hour before surgery, during surgery, and up to 8-24 hours after surgery.

SUMMARY:
The goal of this observational study is to determine the incidence of perioperative cerebral desaturation in neonates undergoing surgery for congenital malformations. The main questions it aims to answer are:

1. The perioperative factors associated with occurrence of cerebral desaturation
2. The association between perioperative cerebral desaturation, perioperative/hospital outcomes, and physiological conditions.

Participants will undergo Near-infrared spectroscopy (NIRS) and electroencephalogram (EEG) monitoring for one hour before surgery, during surgery, and up to 24 hours after surgery.

DETAILED DESCRIPTION:
The NIRS EEG sensors will be placed about an hour before surgery. The recording will start once sensors are placed, continue throughout the duration of surgery, and end 8-24 hours after end of surgery. Sensors will be removed at the end of recording. No additional anesthesia and/or sedation will be required for the preoperative and postoperative recordings. The EEG and NIRS monitors will be blinded to clinical staff. EEG and NIRS monitoring will not prolong anesthesia or the duration of the surgical repair, and should not interfere with routine patient care. NIRS and EEG data will be downloaded from the monitors at the end of recording for analysis.

Medical record review will be conducted at 100 days postop or hospital discharge (whichever is sooner). The information below will be extracted:

* Respiratory record
* Post-op recovery, ICU, and discharge records
* Cardiac and Neurologic records
* Neurologic test such as radiology and lab tests
* Mortality status

ELIGIBILITY:
Inclusion Criteria:

1. Infants ≤ 60 weeks post-menstrual age on day of surgery.
2. Neonatal surgery for congenital abdominal/gastrointestinal malformations (diaphragmatic hernia, gastroschisis, omphalocele, intestinal atresia, Hirschsprung's disease, imperforate anus, necrotizing enterocolitis), congenital cystic adenomatoid/pulmonary airway malformation (CCAM/CPAM), esophageal/tracheoesophageal fistula (EF/TEF), and spinal malformations (myelomeningocele, sacrococcygeal teratoma).
3. The same patient may be enrolled multiple times for repeat or different procedures that meet the above criteria. These subjects will be counted more than once towards the enrollment goal.
4. Parental/guardian permission.

Exclusion Criteria:

1) Patients with hydrocephalus limiting frontal-parietal brain volume, interventricular hemorrhage (grades 3 or 4), malformation or cerebral infarction of frontal-parietal brain.

Max Age: 60 Weeks | Sex: All
Age Groups: Child
Study Population: Infant subjects ≤ 60 weeks post-menstrual age who are undergoing surgery for congenital malformat
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with perioperative cerebral desaturation | 24 hours
  The incidence of cerebral desaturation in participants will be assessed by the Near-infrared Spectroscopy (NIRS) data recording of <70% and/or >10% decrease from baseline for > 3 minutes

SECONDARY OUTCOMES:
Isoelectric EEG | up to 24 hours
  Determined by EEG amplitude ≤ 10mV for ≥ 2 secs
Perioperative outcomes | up to 100 days
  Medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Ian Yuan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (15):
- United States (4):
  - Children's Hospital at Montefiore/Albert Einstein College of Medicine, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
- Australia (2):
  - Perth Children's Hospital, Nedlands
  - Royal Children's Hospital, Parkville
- Hospital das Clínicas, Faculdade de Medicina, Universidade de São Paulo, São Paulo, Brazil
- China (4):
  - Guangzhou women and children's medical center, Guangzhou
  - Shanghai Children's Medical Center, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - West China Hospital and West China Second University Hospital, Sichuan
- Centre Hospitalier Universitaire de Bordeaux, Hopital des enfants, Bordeaux, France
- India (2):
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Christian Medical College Hospital, Vellore
- Great Ormond Street Hospital for Children, London, United Kingdom

REFERENCES:
- [Background] CDC. https://www.cdc.gov/ncbddd/birthdefects/data.html. Accessed April 13, 2021.
- [Background] Bonasso PC, Dassinger MS, Ryan ML, Gowen MS, Burford JM, Smith SD. 24-hour and 30-day perioperative mortality in pediatric surgery. J Pediatr Surg. 2019 Apr;54(4):628-630. doi: 10.1016/j.jpedsurg.2018.06.026. Epub 2018 Jun 25. PMID 30017066
- [Background] Laing S, Walker K, Ungerer J, Badawi N, Spence K. Early development of children with major birth defects requiring newborn surgery. J Paediatr Child Health. 2011 Mar;47(3):140-7. doi: 10.1111/j.1440-1754.2010.01902.x. Epub 2010 Nov 21. PMID 21091587
- [Background] Stolwijk LJ, Lemmers PM, Harmsen M, Groenendaal F, de Vries LS, van der Zee DC, Benders MJ, van Herwaarden-Lindeboom MY. Neurodevelopmental Outcomes After Neonatal Surgery for Major Noncardiac Anomalies. Pediatrics. 2016 Feb;137(2):e20151728. doi: 10.1542/peds.2015-1728. Epub 2016 Jan 12. PMID 26759411
- [Background] Tusor N, Benders MJ, Counsell SJ, Nongena P, Ederies MA, Falconer S, Chew A, Gonzalez-Cinca N, Hajnal JV, Gangadharan S, Chatzi V, Kersbergen KJ, Kennea N, Azzopardi DV, Edwards AD. Punctate White Matter Lesions Associated With Altered Brain Development And Adverse Motor Outcome In Preterm Infants. Sci Rep. 2017 Oct 16;7(1):13250. doi: 10.1038/s41598-017-13753-x. PMID 29038505
- [Background] Stolwijk LJ, Keunen K, de Vries LS, Groenendaal F, van der Zee DC, van Herwaarden MYA, Lemmers PMA, Benders MJNL. Neonatal Surgery for Noncardiac Congenital Anomalies: Neonates at Risk of Brain Injury. J Pediatr. 2017 Mar;182:335-341.e1. doi: 10.1016/j.jpeds.2016.11.080. Epub 2016 Dec 30. PMID 28043688
- [Background] Sood ED, Benzaquen JS, Davies RR, Woodford E, Pizarro C. Predictive value of perioperative near-infrared spectroscopy for neurodevelopmental outcomes after cardiac surgery in infancy. J Thorac Cardiovasc Surg. 2013 Feb;145(2):438-445.e1; discussion 444-5. doi: 10.1016/j.jtcvs.2012.10.033. Epub 2012 Dec 6. PMID 23219333
- [Background] Hoffman GM, Brosig CL, Mussatto KA, Tweddell JS, Ghanayem NS. Perioperative cerebral oxygen saturation in neonates with hypoplastic left heart syndrome and childhood neurodevelopmental outcome. J Thorac Cardiovasc Surg. 2013 Nov;146(5):1153-64. doi: 10.1016/j.jtcvs.2012.12.060. Epub 2013 Jan 12. PMID 23317941
- [Background] Vida VL, Tessari C, Cristante A, Nori R, Pittarello D, Ori C, Cogo PE, Perissinotto E, Stellin G. The Role of Regional Oxygen Saturation Using Near-Infrared Spectroscopy and Blood Lactate Levels as Early Predictors of Outcome After Pediatric Cardiac Surgery. Can J Cardiol. 2016 Aug;32(8):970-7. doi: 10.1016/j.cjca.2015.09.024. Epub 2015 Oct 22. PMID 26868838
- [Background] Danzer E, Hoffman C, D'Agostino JA, Gerdes M, Bernbaum J, Antiel RM, Rintoul NE, Herkert LM, Flake AW, Adzick NS, Hedrick HL. Neurodevelopmental outcomes at 5years of age in congenital diaphragmatic hernia. J Pediatr Surg. 2017 Mar;52(3):437-443. doi: 10.1016/j.jpedsurg.2016.08.008. Epub 2016 Aug 30. PMID 27622588
- [Background] Birthdefects C. https://www.cdc.gov/ncbddd/birthdefects/data.html. Published 2021. Accessed April 21, 2021.
- [Background] Escobar MA Jr, Caty MG. Complications in neonatal surgery. Semin Pediatr Surg. 2016 Dec;25(6):347-370. doi: 10.1053/j.sempedsurg.2016.10.005. Epub 2016 Nov 1. PMID 27989360
- [Background] Andropoulos DB, Ahmad HB, Haq T, Brady K, Stayer SA, Meador MR, Hunter JV, Rivera C, Voigt RG, Turcich M, He CQ, Shekerdemian LS, Dickerson HA, Fraser CD, Dean McKenzie E, Heinle JS, Blaine Easley R. The association between brain injury, perioperative anesthetic exposure, and 12-month neurodevelopmental outcomes after neonatal cardiac surgery: a retrospective cohort study. Paediatr Anaesth. 2014 Mar;24(3):266-74. doi: 10.1111/pan.12350. PMID 24467569
- [Background] Mahle WT, Tavani F, Zimmerman RA, Nicolson SC, Galli KK, Gaynor JW, Clancy RR, Montenegro LM, Spray TL, Chiavacci RM, Wernovsky G, Kurth CD. An MRI study of neurological injury before and after congenital heart surgery. Circulation. 2002 Sep 24;106(12 Suppl 1):I109-14. PMID 12354718
- [Background] Olbrecht VA, Skowno J, Marchesini V, Ding L, Jiang Y, Ward CG, Yu G, Liu H, Schurink B, Vutskits L, de Graaff JC, McGowan FX Jr, von Ungern-Sternberg BS, Kurth CD, Davidson A. An International, Multicenter, Observational Study of Cerebral Oxygenation during Infant and Neonatal Anesthesia. Anesthesiology. 2018 Jan;128(1):85-96. doi: 10.1097/ALN.0000000000001920. PMID 29019815
- [Background] Dent CL, Spaeth JP, Jones BV, Schwartz SM, Glauser TA, Hallinan B, Pearl JM, Khoury PR, Kurth CD. Brain magnetic resonance imaging abnormalities after the Norwood procedure using regional cerebral perfusion. J Thorac Cardiovasc Surg. 2006 Jan;131(1):190-7. doi: 10.1016/j.jtcvs.2005.10.003. PMID 16399311 (Retraction: PMID 16736557 J Thorac Cardiovasc Surg. 2006 Jun;131(6):1226)
- [Background] Suemori T, Skowno J, Horton S, Bottrell S, Butt W, Davidson AJ. Cerebral oxygen saturation and tissue hemoglobin concentration as predictive markers of early postoperative outcomes after pediatric cardiac surgery. Paediatr Anaesth. 2016 Feb;26(2):182-9. doi: 10.1111/pan.12800. Epub 2015 Dec 1. PMID 26619804
- [Background] Kurth CD, Levy WJ, McCann J. Near-infrared spectroscopy cerebral oxygen saturation thresholds for hypoxia-ischemia in piglets. J Cereb Blood Flow Metab. 2002 Mar;22(3):335-41. doi: 10.1097/00004647-200203000-00011. PMID 11891439
- [Background] Yuan I, Xu T, Kurth CD. Using Electroencephalography (EEG) to Guide Propofol and Sevoflurane Dosing in Pediatric Anesthesia. Anesthesiol Clin. 2020 Sep;38(3):709-725. doi: 10.1016/j.anclin.2020.06.007. PMID 32792193
- [Background] Yuan I, Olbrecht VA, Mensinger JL, Zhang B, Davidson AJ, von Ungern-Sternberg BS, Skowno J, Lian Q, Song X, Zhao P, Zhang J, Zhang M, Zuo Y, de Graaff JC, Vutskits L, Szmuk P, Kurth CD. Statistical Analysis Plan for "An international multicenter study of isoelectric electroencephalography events in infants and young children during anesthesia for surgery". Paediatr Anaesth. 2019 Mar;29(3):243-249. doi: 10.1111/pan.13589. PMID 30664323